CLINICAL TRIAL: NCT01162772
Title: Influence of a Modern Oral Anti-diabetic Medication on Endothelial Dysfunction and Cardiovascular Risk in Diabetic Women and Men: Gender Aspects
Brief Title: Influence of DPP-4 on Inflammatory Parameters in Diabetics: Gender Aspects
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Jeanette Strametz-Juranek, MD, Division of Cardiology
Other Study IDs: 575/2008
Record Dates: First submitted 2010-07-13; First posted 2010-07-15 (Estimated); Last update posted 2010-07-16 (Estimated); Status verified 2010-07

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Risk; Endothelial Dysfunction
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Female Diabetics: female, 25-75 years old, no pregnancy, with/out Hormone replacement therapy T2DM, HbA1c > 7% with metformin mono-therapy
- Male diabetics: 25-75 years, T2DM, HbA1c > 7% with metformin mono-therapy

SUMMARY:
Cardiovascular events are the most common cause for death in type 2 diabetes mellitus (T2DM) patients. Male diabetics have a 2 to 3 fold risk for cardiovascular disease (CVD) whereas female diabetes patients have a 3 to 7 fold risk for suffering from a CVD.

Endothelial dysfunction (ED) plays a central role in the development of atherosclerotic lesions. Moreover, ED represents an important diagnostic and prognostic parameter to estimate the cardiovascular risk in an early state. Experimental and clinical studies indicate that T2DM is closely associated with ED, which may be the consequence of a reduced bioactivity of nitric oxide (NO).

The success of diabetes therapy is monitored by the long-term parameter HbA1c. However, only two thirds of all patients with T2DM in the USA and Europe find themselves in the recommended HbA1c span (6.5-7.0 %). Consequently, oral anti-diabetic medication needs permanent adjustment and intensification in order to delaying the progress of T2DM.

Recently, two peptide hormones with insulinotropic effects were identified. These hormones, glucagon-like peptide 1 (GLP-1) and glucose-dependent insulinotropic polypeptide (GIP), are secreted by the gastrointestinal tract after exposure to glucose in nutrition. Physiological effects are increased insulin secretion, inhibition of glucagon secretion and reduction of body weight. Furthermore, these incretins are reduced in patients with impaired glucose tolerance. Thus, the therapeutic approach lies within the elevation of GLP-1 and GIP by preventing their degradation through the enzyme DPP-4 (dipeptidylpeptidase 4).

Thereby, the so-called gliptins inhibit the DPP-4 enzymes. Best results in HbA1c reduction were achieved when gliptins were combined with metformin, glimepiride or pioglitazone.

In this study, patients with T2DM, who are taking metformin as first line medication but do not achieve a HbA1c below 7.0 %, will routinely get an add-on therapy with gliptins (Vildagliptin or Sitagliptin) as second line therapy according to the guidelines of the Österreichische Diabetes Gesellschaft (ÖDG) prescribed by a medical doctor not involved in this study. This medication is a ÖDG standard therapy in T2DM, which patients receive anyway despite this study. Therefore, the therapy with gliptins is not a study medication and is not influenced by the study either. Only patients, who will meet the inclusion criteria of the study and voluntarily participate in the study, will be investigated.

DETAILED DESCRIPTION:
The World Health Organization (WHO) estimates that more than 180 million people worldwide have diabetes. This number is likely to more than double by 2030. Further, the WHO proclaims that diabetes causes about 5 % of all deaths globally each year. Cardiovascular events are the most common cause for death in T2DM patients . According to the VERONA study, which observed 6000 T2DM patients over 10 years, 44 % of all deaths were caused by CVD, primarily heart attack and stroke . Interesting is the fact that male diabetics have a 2 to 3 fold risk for CVD whereas female T2DM patients have a 3 to 7 fold risk for suffering a cardiovascular event although there is no satisfying explanation for this phenomenon.

CVD is caused by atherosclerosis, a condition arising from ED. Hence, ED represents an important diagnostic and prognostic parameter to estimate the cardiovascular risk in a very early state. Such ED is frequently caused by a reduced bioactivity of NO. This molecule is synthesized in endothelial cells by oxidation of L-arginine in a reaction catalyzed by the endothelial nitric oxide synthase . NO is able to protect the vessel wall due to its vasodilatating, anti-adhesive and anti-proliferative activities. Experimental and clinical studies demonstrate that T2DM is closely associated with ED, which may be the consequence of a reduced bioactivity of NO. Central mechanisms explaining this defect in T2DM are the inactivation of NO by reactive oxygen species, the reduction in the amounts of co-factors necessary for NO-synthesis, such as biopterin and NADPH, as well as the inhibition of endothelial NO-synthase by phosphorylation (protein kinase C) and O-glycosylation (hexosamine pathway) .

Endostatin (ENST), an anti-angiogenetic factor, blocks endothelial cell proliferation and migration, induces endothelial cell apoptosis and inhibits thereby angiogenesis . Basal plasma levels of ENST are higher in T2DM patients and thus may be the missing link to explain the inactivation of NO as pro-angiogenetic factor in the process of atherosclerosis.

In T2DM, the high glucose load in the blood leads to swelling of the basement membrane and thus to microangiopathy. This favors the genesis of hypertension due to glomerulosclerosis. Eventually, three factors promote the increased risk for heart attack and stroke:

1. Hypertension
2. Increase of VLDL (due to low insulin levels)
3. and elevated clotting disposition (due to hyperglycemia induced production of fibrinogen, coagulation factor V and VIII) .

One of the difficulties in T2DM is the coexistence of polyneuropathy. As a result symptoms of angina pectoris under stress are painless so that silent infarcts are frequent and often the end point in the CVD progress . Thus, the most important aim in T2DM therapy is the prevention of secondary complications such as CVD. Therefore, the exact adjustment of blood glucose (monitored by HbA1c) plays a pivotal role in prevention. Unfortunately, only two thirds of all patients with T2DM in the USA and Europe find themselves in the recommended HbA1c span (6.5-7.0 %). Consequently, oral anti-diabetic medication needs permanent adjustment and intensification to delay the progress of T2DM. However, metformin and sulfonylurea derail the optimal treatment because of unwanted side effects, especially hypoglycemia and weight gain.

Recently, two peptide hormones, GLP-1 and GIP, with insulinotropic effects were identified. These so-called incretins are secreted by the gastrointestinal tract after exposure to glucose in nutrition. Physiological effects result in

* increased insulin secretion
* inhibition of glucagon secretion
* and reduction of body weight. It has been observed that incretin levels are reduced in patients with impaired glucose tolerance. Thus, the therapeutic approach lies within the elevation of GLP-1 and GIP by preventing their degradation through the enzyme DPP-4 (dipeptidylpeptidase 4), the so-called gliptins that inhibit the DPP-4 enzymes.

Best results in HbA1c reduction were achieved when gliptins were combined with metformin, glimepiride or pioglitazone .

In this study, patients with T2DM, who are taking metformin as first line medication but do not achieve a HbA1c below 7.0 % and with an intolerance against sulfonylurea (hypoglycemia during the night) and glitazones (obesity, weight gain and ankle edema), will routinely get an add-on therapy with gliptins (Vildagliptin or Sitagliptin) as second line therapy according to the guidelines of the Österreichische Diabetes Gesellschaft (ÖDG) prescribed by a medical doctor not involved in this study. This medication is a ÖDG standard therapy in T2DM, which patients receive anyway despite this study. Therefore, the therapy with gliptins is not a study medication and is not influenced by the study either. Only patients, who will meet the inclusion criteria of the study and voluntarily participate in the study, will be investigated.

Rationale of the study

This study aims to investigate the effects of a modern oral anti-diabetic medication according to the guidelines of the ÖDG on ED. A special focus will be put on the outcome between female and male patients to elucidate the different effects of the drugs on inflammatory parameters in women and men.

The following parameters will be measured:

* Catecholamine (norepinephrine, dopamine, epinephrine) Catecholamines are released by the adrenal gland in situations of stress such as psychological stress, physical stress or low blood sugar levels . They are water-soluble and 50 % bound to plasma proteins. The three major catecholamines that circulate in the blood are epinephrine, norepinephrine and dopamine. They are mainly produced from the adrenal medulla and the postganglionic fibers of the sympathetic nervous system. The measurement of the catecholamines serves as control parameter for the applied stress situations.
* ENST ENST, a 20-kDa C-terminal fragment derived from type XVIII collagen, is an endogenous protein that blocks the formation of blood vessels. It inhibits endothelial cell proliferation, migration and angiogenesis. There is evidence for several functions of neovascularisation in plaque growth that maintain perfusion beyond limits of diffusion from the artery lumen and outer adventitial vasa vasorum, deposit pro-atherogenic plasma molecules, recruit immune cells and progenitors, and promote intraplaque hemorrhage . ENST, as an angiostatic factor, might be the weapon of choice to battle these effects.
* BNP Brain natriuretic peptide (BNP) is a 32-amino acid peptide . It is synthesized predominantly in the left ventricle of the heart as the 108-amino acid pro-hormone preproBNP ( -BNP) . The hormone is a potent vasodilator and a natriuretic factor regulating salt and water homeostasis. BNP is stored in the human cardiac tissue mainly as BNP-32 with a lesser amount of the precursor preproBNP. The circulating plasma forms of BNP are BNP-32 and the NH2-terminal portion proBNP (Nt-proBNP) . Increased secretion of BNP and Nt-proBNP occurs mainly with increased tension in the ventricular walls, decreased oxygen supply, acute myocardial infarction, chronic cardiac heart failure, and in hypertrophy of the heart . The Nt-proBNP level was shown to be significantly elevated in the cohort of patients with T2DM. Taken together, both BNP and Nt-proBNP serve as sensitive markers of CVD .
* Intima-media thickness (by carotid-ultrasound) IMT is a measurement of the thickness of artery walls, usually by external ultrasound, to detect the presence and to track the progression of atherosclerotic lesions. Cross-sectional associations between common carotid artery IMT and cardiovascular risk factors have been demonstrated in several studies .
* Heart rate
* Blood pressure
* ECG

ELIGIBILITY:
Inclusion Criteria:

* patients with T2DM
* metformin therapy
* HbA1c < 7%
* 25 - 69 years

Exclusion Criteria:

* pregnant women
* untreated thyroid dysfunction
* renal insufficiency (creatinine clearance < 60 ml/min)
* unstable coronary heart disease
* NYHA III or IV
* severe hepatic dysfunction except steatosis (GOT and GPT three times higher than ULN)
* patients undergoing cortisone therapy
* condition post stroke within the last 6 months

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: In this study 40 female and 40 male subjects with T2DM, who take metformin as an oral anti-diabetic mono therapy according to the guidelines of the ÖDG.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Endostatin | Baseline
  ENST, a 20-kDa C-terminal fragment derived from type XVIII collagen, is an endogenous protein that blocks the formation of blood vessels. It inhibits endothelial cell proliferation, migration and angiogenesis. There is evidence for several functions of neovascularisation in plaque growth that maintain perfusion beyond limits of diffusion from the artery lumen and outer adventitial vasa vasorum, deposit pro-atherogenic plasma molecules, recruit immune cells and progenitors, and promote intraplaque hemorrhage . ENST, as an angiostatic factor, might be the weapon of choice to battle these effects
catecholamine | baseline
  Catecholamines are released by the adrenal gland in situations of stress such as psychological stress, physical stress or low blood sugar levels . They are water-soluble and 50 % bound to plasma proteins. The three major catecholamines that circulate in the blood are epinephrine, norepinephrine and dopamine. They are mainly produced from the adrenal medulla and the postganglionic fibers of the sympathetic nervous system. The measurement of the catecholamines serves as control parameter for the applied stress situations.
Endostatin | after 6 months
catecholamine | after 6 months

SECONDARY OUTCOMES:
Brain natriuretic peptide | baseline
  Brain natriuretic peptide (BNP), a 32-amino acid peptide synthesized predominantly in the left ventricle of the heart as the 108-amino acid prohormone, is a potent vasodilator and a natriuretic factor regulating salt and water homeostasis.. Increased secretion of BNP and Nt-proBNP occurs mainly with increased tension in the ventricular walls, decreased oxygen supply, acute myocardial infarction, chronic cardiac heart failure, and in hypertrophy of the heart.
  The Nt-proBNP level was shown to be significantly elevated in the cohort of patients with diabetes.
Intima media thickness | baseline
  IMT is a measurement of the thickness of artery walls, usually by external ultrasound, to detect the presence and to track the progression of atherosclerotic lesions. Cross-sectional associations between common carotid artery IMT and cardiovascular risk factors have been demonstrated in several studies
Sex hormones | baseline
  Total testosterone concentrations in the low-normal range predict diabetes and the development of the metabolic syndrome as defined by the NCEP in middle-aged men, independently of BMI and other factors related to insulin resistance. Hyperandrogenicity in women is closely associated with insulin resistance and presents a risk factor for CVD and T2DM. Hormone replacement therapy improves glucose homeostasis and lipoprotein profile. T2DM abolishes the female-gender related differences in the risk of CVD, and diabetic women have rates of ischemic heart disease mortality approaching those of men.
Plasminogen Activator inhibitor-1 | baseline
  Plasminogen activator inhibitor 1 (PAI-1) is the primary physiological inhibitor of plasminogen activation in vivo. Circulating PAI-1 levels are elevated in patients with coronary heart disease and may play an important role in the development of atherothrombosis by decreasing fibrin degradation. Increased PAI-1 expression can also directly influence vessel wall remodelling. The insulin resistance syndrome, which is characterized partly by obesity with visceral fat accumulation, is considered as a major regulator of PAI-1 expression
Adrenomedullin | baseline
  Adrenomedullin (AM) has multi-functional properties, of which the vasodilatory hypotensive effect is the most characteristic. AM secretion, especially in cardiovascular tissues, is regulated mainly by mechanical stressors (shear stress, inflammatory and metabolic factors). Elevation of plasma AM due to overproduction in response to one or more of these stimuli in pathological conditions may explain the raised plasma AM levels present in cardiovascular diseases such as myocardial infarction, hypertension, stroke and diabetes mellitus
Ultra sensitive C-reactive protein | baseline
  Endothelial activation and acute-phase reaction correlate with insulin resistance and obesity in T2DM patients. Prospective studies have shown that ultra sensitive C-reactive protein (usCRP) can be used to predict risk of future cardiovascular events
Asymmetric dimethylarginine | baseline
  Increased plasma concentration of asymmetric dimethylarginine (ADMA), an endogenous inhibitor of nitric oxide synthase, is associated with endothelial dysfunction, insulin resistance, and atherosclerosis and might, thus, serve as a marker for cardiovascular morbidity. In T2DM, the release and/or bioavailibility of nitric oxide are diminished. This endogenous nitric oxide synthase inhibitor, ADMA, has recently emerged as a key factor in nitric oxide biosynthesis.
Adiponectin | baselie and after 6 months
  Adiponectin is a hormone secreted by visceral adipose tissue beside others like leptin, angiotensin and resistin and exhibits antiinflammatory and insulin-sensitizing properties. Low plasma adiponectin concentrations have been suggested to promote atherosclerosis and have been found to be associated with early CVD onset and multiple atherosclerotic lesions in coronary arteries. Thus, adiponectin concentrations may influence risk of CVD and might serve as one of the screening tests facilitating early intervention
Apelin | baseline
  Apelin, a newly discovered adipocytokine and inotropic agent, is produced by white adipose tissue and is also expressed in the kidney and heart. Increasing evidence suggests a role for apelin in the pathology of the cardiovascular system. Plasma apelin is reduced in newly diagnosed and untreated patients with T2DM. Regulation of circulating apelin and adiponectin seems to be in the same manner in patients with T2DM. Dysregulation of apelin might be involved in the mechanism of establishment of overt diabetes mellitus as well as associated atherosclerotic complications.
Homeostasis model assessment-estimated insulin resistance | baseline
  The Homeostasis model assessment of insulin resistance (HOMA-IR) is calculated by multiplying fasting insulin (μU/ml) and fasting blood sugar (mg/dl) divided through 19 (Version 1.2. vom 08.12.2008)
  . A HOMA-IR below 1 is regarded as normal whereas a value over 2 is a hint for insulin resistance. The HOMA-IR has been suggested as a method to assess insulin resistance and secretion from the fasting glucose and insulin concentrations. T2DM is characterized by high HOMA IR. The HOMA-IR is an independent predictor of CVD in T2DM.
Brain natriuretic peptide | after 6 months
Intima media thickness | after 6 months
Sex hormones | after 6 months
Plasminogen Activator inhibitor-1 | after 6 months
Adrenomedullin | after 6 months
Ultra sensitive C-reactive protein | after 6 months
Asymmetric dimethylarginine | after 6 months
Apelin | after 6 moths
Homeostasis model assessment-estimated insulin resistance | after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeanette Strametz-Juranek, MD, Principal Investigator — MUV, Department of Internal Medicine II, Division of Cardiology; Alexandra Kautzky-Willer, MD, Principal Investigator — MUV, Department of Medicine III, Division of Endocrinology
Locations (1):
- Medical University of Viemma, Vienna, Austria